CLINICAL TRIAL: NCT03081442
Title: Benefits of Use of 600 Microgram Misoprostol Vaginally Prior To Insertion Of An Intrauterine Device in Patients With Cesarean Scar: A Randomized Controlled Trial
Brief Title: Vaginal Misoprostol Before IUD Insertion in Women With Cesarean Scar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 159
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Contraceptive Device; Complications
MeSH Terms: interventions — Misoprostol; Intrauterine Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol group (Active Comparator): Sixty women received 600 micrograms of misoprostol vaginally as deep as possible six hours before IUD insertion.
  Interventions: Drug: Misoprostol; Device: Intrauterine contraceptive device IUCD
- placebo group (Placebo Comparator): Sixty women received the placebo vaginally six hours before IUD insertion. Placebo is the same in size, color and shape to misoprostol.
  Interventions: Device: Intrauterine contraceptive device IUCD

INTERVENTIONS:
Drug: Misoprostol — 600 micrograms of misoprostol vaginally as deep as possible six hours before IUD insertion
  Other Names: cytotec
  Arms: Misoprostol group
Device: Intrauterine contraceptive device IUCD — bimanual examination. The cervix was exposed by introducing a vaginal speculum, the cervix and vaginal vault were cleaned with povidone- iodine solution.
  The Next step was to sound The IUD was folded into the insertion tube immediately prior to insertion. The cervix was grasped with a tenaculum, and gently pulled downward The insertion tube was advanced into the uterus to the correct depth as marked on the tube by a sliding plastic flange.
  The outer sheath of the insert was withdrawn ashort distance to release the arms of the T and was then gently pushed inward again to elevate the opened T against the fundus of uterus .
  Other Names: TCu-380A®,Pregna International Ltd, India

SUMMARY:
Groups of study:

120 candidates for Cu T 380A IUD insertion were enrolled in the study. They were divided into two groups: Group 1: Sixty women received 600 micrograms of misoprostol vaginally as deep as possible six hours before IUD insertion.

Group 2: Sixty women received the placebo vaginally. The placebo and misoprostol were put in 120 numbered closed envelopes according to the table of random numbers and an envelope was allocated to each patient accordingly.

Methodology:

All patients were subjected to the following:

(i) Complete history taking (ii) Proper counseling: (iv) Examination: (v) 600ug misoprostol (3tablets Misotac®, ( Sigma Pharmaceutical Industries, Egypt )or placebo were administered Vaginally as deep as possible 6 hours before insertion of the IUD by gynecologist .

(vi) Insertion of IUD: (TCu-380A®,Pregna International Ltd, India ) After full history taken , Proper counseling, Informed consent is taken from each patients, examination ( general , abdominal and pelvic )to exclude any pathology .

A careful bimanual examination was done prior to IUD insertion. The cervix was exposed by introducing a vaginal speculum, the cervix and vaginal vault were cleaned with povidone- iodine solution.

The Next step was to sound and measure the depth of the uterus. The IUD was folded into the insertion tube immediately prior to insertion. The cervix was grasped with a tenaculum, and gently pulled downward to straighten the angle of flection.

The insertion tube was advanced into the uterus to the correct depth as marked on the tube by a sliding plastic flange.

The outer sheath of the insert was withdrawn a short distance to release the arms of the T and was then gently pushed inward again to elevate the opened T against the fundus of uterus .

The inserter tube was then removed. Then strings were cut to project about 2-4 cm from the external cervical os.

DETAILED DESCRIPTION:
Groups of study:

120 candidates for Cu T 380A IUD insertion were enrolled in the study. They were divided into two groups: Group 1: Sixty women received 600 micrograms of misoprostol vaginally as deep as possible six hours before IUD insertion.

Group 2: Sixty women received the placebo vaginally. The placebo and misoprostol were put in 120 numbered closed envelopes according to the table of random numbers and an envelope was allocated to each patient accordingly.

Methods of randomization:

To insure that everyone had an equal chance of participation, randomization was guided by table of random numbers using computer generated system(SPSS: windous version8) (SPSS Inc., Chicago, USA) double blinding technique was used thus; the investigator and the patient didn't know the group to which the patient was allocated.

Methodology:

All patients were subjected to the following:

(i) Complete history taking:

* Full history taking.
* Obstetric history.
* Menstrual history.
* Medical history. Data were collected in a special form for each patient. (ii) Proper counseling: Proper counseling of each patient about different types of IUDs, the advantage and side effects of each type, explanation of the menstrual pattern changes, assuring the patient that these changes are very common and that it will disappear after a period of time after insertion.

(iii) Consent: Informed consent is taken from each patients . (iv) Examination:

1. General examination.
2. Abdominal examination.
3. Pelvic examination to exclude pelvic pathology .

   (v) 600ug misoprostol (3tablets Misotac®, ( Sigma Pharmaceutical Industries, Egypt )or placebo ( stugeron®, Mina Pharm. under licence Janssen Pharmaceutica, Egypt ) were administered Vaginally as deep as possible 6 hours before insertion of the IUD by gynecologist .

   (vi) Insertion of IUD: (TCu-380A®,Pregna International Ltd, India ) After full history taken , Proper counseling, Informed consent is taken from each patients, examination ( general , abdominal and pelvic )to exclude any pathology .

   A careful bimanual examination was done prior to IUD insertion. The cervix was exposed by introducing a vaginal speculum, the cervix and vaginal vault were cleaned with povidone- iodine solution.

   The Next step was to sound and measure the depth of the uterus. The IUD was folded into the insertion tube immediately prior to insertion. The cervix was grasped with a tenaculum, and gently pulled downward to straighten the angle of flection.

   The insertion tube was advanced into the uterus to the correct depth as marked on the tube by a sliding plastic flange.

   The outer sheath of the insert was withdrawn ashort distance to release the arms of the T and was then gently pushed inward again to elevate the opened T against the fundus of uterus .

   The inserter tube was then removed. Then strings were cut to project about 2-4 cm from the external cervical os.

   Post insertion instructions:

   Palpation of strings should be performed monthly by the patient to verify continuing presence of the IUD after each menstrual flow. Caution the patient that the first 2 menses are typically heavier.

ELIGIBILITY:
Inclusion Criteria:

* Women with previous cesarean section and with no previous vaginal delivery attending outpatient clinic for IUD insertion

Exclusion Criteria:

1. contraindications for misoprostol use (pregnancy and prostaglandin allergy).
2. contraindications for IUD use (gynecologic malignancy, pelvic inflammatory disease and unexplained vaginal bleeding).
3. previous vaginal delivery. And (4) medical disorders as diabetes, hypertension and bleeding tendency .

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Pain score | At time of insertion
  Pain scores were measured by Visual analogue scale (VAS) consists of 10 cm horizontal straight line with 2 ends At 0 end there was no pain and at 10 there was a severe pain

SECONDARY OUTCOMES:
Difficulty of insertion of IUD in both groups | At time of insertion
  Difficulty of IUD insertion was measured by a 10-point scale, on which 0 represented an extremely easy, and 10 an extremely difficult insertion
side effects | from time of administration till insertion
  abdominal cramps, headache, nausea, diarrhea and fever

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No